CLINICAL TRIAL: NCT00553865
Title: A 8-Week, Randomized, Double-blind, Parallel Designed, Phase II Multi-center Clinical Trial to Evaluate the Antihypertensive Efficacy and the Safety of OJP-2028 Tablets in Patients With the Uncomplicated Essential Hypertension
Brief Title: Clinical Trial to Evaluate the Efficacy and the Safety of Antihypertensive Tablets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OJP-2028-II
Record Dates: First submitted 2007-11-03; First posted 2007-11-06 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2014-09

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Experimental): OJP-2028 1mg/day
  Interventions: Drug: OJP-2028
- Group 2 (Experimental): OJP-2028 2mg/day
  Interventions: Drug: OJP-2028
- Group 3 (Experimental): OJP-2028 4mg/day
  Interventions: Drug: OJP-2028
- Group 4 (Placebo Comparator): Placebo
  Interventions: Drug: OJP-2028
- Group 5 (Other): Reference drug
  Interventions: Drug: OJP-2028

INTERVENTIONS:
Drug: OJP-2028 — Experimental: 1mg/day, 2mg/day, 4mg/day for 8 weeks. Placebo Comparator: Placebo.day for 8 weeks. Reference group(Group 5): Reference Drug/day for 8 weeks.

SUMMARY:
The purpose of this study is to determine the optimal dosage of the clinical trial which is evaluating the antihypertensive efficacy and the safety of OJP-2028 tablets in patients with the uncomplicated essential hypertension.

DETAILED DESCRIPTION:
Evaluating the antihypertensive efficacy and the safety of OJP-2028 tablets in patients with the uncomplicated essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women (Age 18-75 years)
2. Uncomplicated essential hypertension: Clinic sitting SiDBP between 90 and 109 mmHg after 2 week placebo run-in period

Exclusion Criteria:

1. Secondary hypertension
2. History and/or signs of cardiovascular complications (eg; myocardial infarction, unstable angina)
3. Pregnancy or lactation
4. Contraindications to the antihypertensive drugs to be used during the treatment period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Average SiDBP Differences of test group vs control group per each dosage by comparison with the baseline. | 8 weeks

SECONDARY OUTCOMES:
Average SiSBP Differences of each group by comparison with the baseline. | 8 weeks
Responder rate of each group by comparison with the baseline. | 8 weeks
Average SiDBP and SiSBP Differences of each group by comparison with the baseline. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: CHEOL HO KIM, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No